CLINICAL TRIAL: NCT07341516
Title: Worldwide Assessment of Deceased Donor Kidney Utilization: Disparities, Temporal Trends, and Outcomes
Brief Title: Worldwide Assessment of Deceased Donor Kidney Utilization
Status: Enrolling by invitation | Type: Observational
Sponsor: Paris Translational Research Center for Organ Transplantation (Other)
Collaborators: Vanderbilt University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: Kidney allocation project
Record Dates: First submitted 2025-12-17; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-12

CONDITIONS: Kidney Failure; Kidney Transplant; Deceased Donor Kidney Transplant
Keywords: kidney transplantation; allocation; deceased donor; organ utilization
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The persistent imbalance between kidney transplant demand and organ availability remains a major global challenge. Optimizing the utilization of kidneys from deceased donors is a critical strategy to expand the donor pool and increase access to transplantation. Previous studies have demonstrated substantial international differences in kidney acceptance and discard practices, with significant potential gains in allograft life-years through optimized utilization. However, major changes in allocation policies, donor characteristics, preservation technologies, and global events such as the COVID-19 pandemic may have altered contemporary utilization patterns. This study aims to characterize international trends in deceased donor kidney utilization, compare allograft survival across countries, and estimate potential transplantable allograft life-years gained through improved utilization practices.

DETAILED DESCRIPTION:
Substantial imbalance between organ demand and availability remains a major challenge in kidney transplantation worldwide. Therefore, expanding the donor pool is a critical priority, and a key strategy is optimizing the utilization of organs from deceased donors. Our previous study (PMID: 31449299) demonstrated significant disparities in kidney acceptance and discard rates between US and France, with US discarding kidneys at nearly twice the rate of France. Simulation modeling suggested that adopting more aggressive, French-based acceptance practices could have prevented 17 435 discarded kidneys in the US over ten years, generating an additional 132 445 allograft life-years.

Since that period the transplantation landscape has evolved substantially. Key developments include major policy reforms such as the 2014 US Kidney Allocation System redesign, increased use of advanced preservation technologies, expanding acceptance of hepatitis C-positive donor organs, substantial growth in donation after circulatory death (DCD), and global disruptions in transplant activity caused by the COVID-19 pandemic.

The impact of these developments on current utilization practices and international disparities remains unknown. Contemporary patterns of deceased donor kidney utilization and discard rates across different allocation systems have not yet been characterized.

This study aims to:

1. Characterize international patterns and temporal trends in deceased donor kidney utilization and discard rates from 2010 to 2025.
2. Compare allograft survival across countries and donor risk profiles.
3. Quantify potential transplantable allograft life-years gained through optimized utilization practices.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive kidneys recovered for the purpose of transplantation from donors deceased from brain death or circulatory death between January 1, 2010 and December 31, 2025

Exclusion Criteria:

* Kidneys offered to transplant centers but never recovered
* Living renal transplants
* Multiorgan transplant recipients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All kidneys recovered for transplantation from deceased donors (brain death or circulatory death) between January 1, 2010, and December 31, 2025, across 10 allocation systems, with sufficient data to calculate the Kidney Donor Risk Index. Recipients of transplants from these donors will also be included for outcome assessment.
Sampling Method: Non-Probability Sample
Enrollment: 300000 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Kidney allograft discard | Day 0
  defined as kidneys recovered for transplantation but not transplanted.

SECONDARY OUTCOMES:
Allograft failure | up to 15 years
  defined as return to dialysis and/or re-transplantation.
Estimated additional allograft life-years achievable | up to 15 years
  through adoption of best practice utilization patterns (simulation based).

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Loupy, MD, PhD, Principal Investigator — Paris Institute for Transplantation and Organ Regeneration, INSERM, UMR-S970, Paris, France; Peter P Reese, MD, PhD, Principal Investigator — Vanderbilt Center for Transplant Science, Vanderbilt University Medical Center, Nashville, TN, USA
Locations (2):
- Vanderbilt Center for Transplant Science, Vanderbilt University Medical Center, Nashville, TN, USA, Nashville, Tennessee, United States
- Paris Institute for Transplantation and Organ Regeneration, INSERM, UMR-S970, Paris, France, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided
The data analyzed during the current study are available on reasonable request including standards for General Data Protection Regulation and Institutional Review Board approval.

REFERENCES:
- [Background] Aubert O, Yoo D, Zielinski D, Cozzi E, Cardillo M, Durr M, Dominguez-Gil B, Coll E, Da Silva MI, Sallinen V, Lemstrom K, Midtvedt K, Ulloa C, Immer F, Weissenbacher A, Vallant N, Basic-Jukic N, Tanabe K, Papatheodoridis G, Menoudakou G, Torres M, Soratti C, Hansen Krogh D, Lefaucheur C, Ferreira G, Silva HT Jr, Hartell D, Forsythe J, Mumford L, Reese PP, Kerbaul F, Jacquelinet C, Vogelaar S, Papalois V, Loupy A. COVID-19 pandemic and worldwide organ transplantation: a population-based study. Lancet Public Health. 2021 Oct;6(10):e709-e719. doi: 10.1016/S2468-2667(21)00200-0. Epub 2021 Aug 30. PMID 34474014
- [Background] Loupy A, Aubert O, Reese PP, Bastien O, Bayer F, Jacquelinet C. Organ procurement and transplantation during the COVID-19 pandemic. Lancet. 2020 May 23;395(10237):e95-e96. doi: 10.1016/S0140-6736(20)31040-0. Epub 2020 May 11. No abstract available. PMID 32407668
- [Background] Ibrahim M, Vece G, Mehew J, Johnson R, Forsythe J, Klassen D, Callaghan C, Stewart D. An international comparison of deceased donor kidney utilization: What can the United States and the United Kingdom learn from each other? Am J Transplant. 2020 May;20(5):1309-1322. doi: 10.1111/ajt.15719. Epub 2019 Dec 21. PMID 31758833
- [Background] Vidgren M, Delorme C, Oniscu GC. Challenges and opportunities in organ donation after circulatory death. J Intern Med. 2025 Feb;297(2):124-140. doi: 10.1111/joim.20051. Epub 2025 Jan 20. PMID 39829342
- [Background] Potluri VS, Goldberg DS, Mohan S, Bloom RD, Sawinski D, Abt PL, Blumberg EA, Parikh CR, Sharpe J, Reddy KR, Molnar MZ, Sise M, Reese PP. National Trends in Utilization and 1-Year Outcomes with Transplantation of HCV-Viremic Kidneys. J Am Soc Nephrol. 2019 Oct;30(10):1939-1951. doi: 10.1681/ASN.2019050462. Epub 2019 Sep 12. PMID 31515244
- [Background] Bowring MG, Shaffer AA, Massie AB, Cameron A, Desai N, Sulkowski M, Garonzik-Wang J, Segev DL. Center-level trends in utilization of HCV-exposed donors for HCV-uninfected kidney and liver transplant recipients in the United States. Am J Transplant. 2019 Aug;19(8):2329-2341. doi: 10.1111/ajt.15355. Epub 2019 Apr 9. PMID 30861279
- [Background] Hosgood SA, Callaghan CJ, Wilson CH, Smith L, Mullings J, Mehew J, Oniscu GC, Phillips BL, Bates L, Nicholson ML. Normothermic machine perfusion versus static cold storage in donation after circulatory death kidney transplantation: a randomized controlled trial. Nat Med. 2023 Jun;29(6):1511-1519. doi: 10.1038/s41591-023-02376-7. Epub 2023 May 25. PMID 37231075
- [Background] Malinoski D, Saunders C, Swain S, Groat T, Wood PR, Reese J, Nelson R, Prinz J, Kishish K, Van De Walker C, Geraghty PJ, Broglio K, Niemann CU. Hypothermia or Machine Perfusion in Kidney Donors. N Engl J Med. 2023 Feb 2;388(5):418-426. doi: 10.1056/NEJMoa2118265. PMID 36724328
- [Background] Moers C, Smits JM, Maathuis MH, Treckmann J, van Gelder F, Napieralski BP, van Kasterop-Kutz M, van der Heide JJ, Squifflet JP, van Heurn E, Kirste GR, Rahmel A, Leuvenink HG, Paul A, Pirenne J, Ploeg RJ. Machine perfusion or cold storage in deceased-donor kidney transplantation. N Engl J Med. 2009 Jan 1;360(1):7-19. doi: 10.1056/NEJMoa0802289. PMID 19118301
- [Background] Stewart DE, Garcia VC, Rosendale JD, Klassen DK, Carrico BJ. Diagnosing the Decades-Long Rise in the Deceased Donor Kidney Discard Rate in the United States. Transplantation. 2017 Mar;101(3):575-587. doi: 10.1097/TP.0000000000001539. PMID 27764031
- [Background] Aubert O, Reese PP, Audry B, Bouatou Y, Raynaud M, Viglietti D, Legendre C, Glotz D, Empana JP, Jouven X, Lefaucheur C, Jacquelinet C, Loupy A. Disparities in Acceptance of Deceased Donor Kidneys Between the United States and France and Estimated Effects of Increased US Acceptance. JAMA Intern Med. 2019 Oct 1;179(10):1365-1374. doi: 10.1001/jamainternmed.2019.2322. PMID 31449299
- See also: Related Info — https://clinicaltrials.gov